CLINICAL TRIAL: NCT02735018
Title: Randomized Double-blind Clinical Trial Comparing the Cardiovascular Effects of Local Anesthesia Solutions Containing 1:100,000 and 1:200,000 of Epinephrine Concentrations
Brief Title: Comparing Cardiovascular Effects of 1:100,000 and 1:200,000 Epinephrine Solutions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Fabio Ritto, DDS, MD, MS, PhD, Program Director, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 496.117
Record Dates: First submitted 2016-03-18; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Cardiovascular Response to Epinephrine
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Epinephrine 1:100,000 (Experimental): Inferior alveolar nerve block with Epinephrine 1:100.000
  Interventions: Drug: Epinephrine 1:100,000
- Epinephrine 1:200,000 (Experimental): Inferior alveolar nerve block with Epinephrine 1:200.000
  Interventions: Drug: Epinephrine 1:200,000

INTERVENTIONS:
Drug: Epinephrine 1:100,000 — Inferior alveolar nerve block with Epinephrine 1:100.000
  Arms: Epinephrine 1:100,000
Drug: Epinephrine 1:200,000 — Inferior alveolar nerve block with Epinephrine 1:200.000
  Arms: Epinephrine 1:200,000

SUMMARY:
The study aim to evaluate systemic response of patients when 2 different concentrations of Epinephrine are injected during inferior alveolar nerve block for wisdom teeth extraction.

ELIGIBILITY:
Inclusion Criteria:

* Class I patients according to the American Society of Anesthesiology (ASA),
* Indication for third molars extraction,
* Similar degree of complexity, according to the classification of Pell and Gregory.

Exclusion Criteria:

* Patients with systemic conditions,
* Patients with known allergy to any component of the anesthetic solution.

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Heart rate | 20 minutes
Blood pressure | 20 minutes
Arterial oxygen saturation, measured with a pulse oximeter device | 20 minutes
Bleeding, evaluated by the surgeon as either: 1) normal or 2) excessive | 20 minutes
Pain, evaluated using a visual analogue scale | After procedure, about 1 hour